CLINICAL TRIAL: NCT00151320
Title: Phase I/II Trial of VELCADE+ CHOP-Rituximab in Patients With Previously Untreated Diffuse Large B Cell or Mantle Cell Non-Hodgkin's Lymphoma
Brief Title: Phase I/II Trial of VELCADE + CHOP-Rituximab in Untreated DLCBL or Mantle Cell NHL
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0309006313
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Results first posted 2017-04-07 (Actual); Last update posted 2018-06-19 (Actual); Status verified 2018-05

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: diffuse large B cell; mantle cell lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Mantle-Cell | interventions — Bortezomib; Rituximab

STUDY DESIGN:
Intervention Model Description: Standard CHOP chemotherapy administered every 21 days (full dose) for six cycles
  Rituximab administered (375 mg/m2) day 1 of each cycle (with usual premedications)
  VELCADE is administered prior to rituximab and CHOP on day 1 of each cycle. The dose of VELCADE will be determined by the dose escalation schedule.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): Standard CHOP chemotherapy administered every 21 days (full dose) for six cycles
  Rituximab administered (375 mg/m2) day 1 of each cycle (with usual premedications)
  VELCADE (Bortezomib) is administered prior to rituximab and CHOP on day 1 of each cycle. The dose of VELCADE will be determined by a dose escalation schedule.
  Interventions: Drug: Bortezomib, CHOP, Rituximab

INTERVENTIONS:
Drug: Bortezomib, CHOP, Rituximab — Standard CHOP chemotherapy administered every 21 days (full dose) for six cycles Rituximab administered (375 mg/m2) day 1 of each cycle (with usual premedications)
  VELCADE (Bortezomib) is administered prior to rituximab and CHOP on day 1 of each cycle. The dose of VELCADE will be determined by the following dose escalation schedule:
  Level Dose/Schedule (-2) 0.7 mg/m2 on day 1 of each cycle (-1) 0.7 mg/m2 on days 1 and 8 (0) 0.7 mg/m2 on days 1 and 4 (+1) 1.0 mg/m2 on days 1 and 4 (+2) 1.3 mg/m2 on days 1 and 4
  Other Names: VELCADE

SUMMARY:
Primary Objective:

To determine the toxicity profile and maximum tolerated dose (MTD) of VELCADE when administered in combination with CHOP + Rituximab to patients with previously untreated diffuse large B cell or mantle cell non-Hodgkin's lymphoma (NHL)

Secondary Objectives:

To assess the response rate (overall and complete), event-free survival and overall survival with VELCADE and CHOP-R in patients with previously untreated diffuse large B cell or mantle cell lymphoma (phase II component)

Treatment:

Standard CHOP chemotherapy administered every 21 days (full dose) for six cycles

Rituximab administered (375 mg/m2) day 1 of each cycle (with usual premedications)

VELCADE is administered prior to rituximab and CHOP on day 1 of each cycle. The dose of VELCADE will be determined by the following dose escalation schedule:

Level Dose/Schedule (-2) 0.7 mg/m2 on day 1 of each cycle (-1) 0.7 mg/m2 on days 1 and 8 (0) 0.7 mg/m2 on days 1 and 4 (+1) 1.0 mg/m2 on days 1 and 4 (+2) 1.3 mg/m2 on days 1 and 4

DETAILED DESCRIPTION:
Standard CHOP chemotherapy administered every 21 days (full dose) for six cycles

Rituximab administered (375 mg/m2) day 1 of each cycle (with usual premedications)

VELCADE is administered prior to rituximab and CHOP on day 1 of each cycle. The dose of VELCADE will be determined by the following dose escalation schedule:

Once completed six cycles of therapy (~18 weeks), patients will be evaluated every 3 months for the first year post treatment, then every 6 months until disease progression or death for years 2 through 5 post treatment. Patients who have disease progression will be contacted every 6 months until death to assess for survival status.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of diffuse large B cell or mantle cell Non-Hodgkin's Lymphoma with characteristic immunophenotypic profiles. For mantle cell: CD5(+), CD19(+) or CD20(+), cyclin D1(+), CD23(-) and CD10(-).
* Patient has not received any prior anti-cancer therapy for lymphoma
* Tumor tissue confirmed to express the CD20 antigen
* Available frozen tumor tissue(rebiopsy if needed)
* Patient has measurable disease as defined by a tumor mass > 1.5 cm
* Patient has Stage II, III, or IV disease
* Age > 18 years
* Absolute granulocyte count > 1000 cells/mm3
* Platelet count > 50,000 cells/mm3
* Creatinine < 2.0 x ULN
* Total bilirubin < 2.0 x ULN

Exclusion Criteria:

* Known central nervous system (CNS) involvement by lymphoma
* Known HIV disease
* Patient is pregnant or nursing
* Patient has had major surgery within the last 3 weeks
* Patient is receiving other investigational drugs
* Known peripheral neuropathy > Grade 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2004-01 (Actual); Primary Completion 2010-04 (Actual); Study Completion 2013-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John P Leonard, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (4):
- United States (4):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Nebraska Medical Center, Omaha, Nebraska
  - Weill Medical College of Cornell University, New York, New York
  - Columbia University College of Physicians and Surgeons, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Standard CHOP chemotherapy administered every 21 days (full dose) for six cycles
  Rituximab administered (375 mg/m2) day 1 of each cycle (with usual premedications)
  VELCADE (Bortezomib) is administered prior to rituximab and CHOP on day 1 of each cycle. The dose of VELCADE will be determined by a dose escalation schedule.
  Bortezomib, CHOP, Rituximab: Standard CHOP chemotherapy administered every 21 days (full dose) for six cycles Rituximab administered (375 mg/m2) day 1 of each cycle (with usual premedications)
  VELCADE (Bortezomib) is administered prior to rituximab and CHOP on day 1 of each cycle. The dose of VELCADE will be determined by the following dose escalation schedule:
  Level Dose/Schedule (-2) 0.7 mg/m2 on day 1 of each cycle (-1) 0.7 mg/m2 on days 1 and 8 (0) 0.7 mg/m2 on days 1 and 4 (+1) 1.0 mg/m2 on days 1 and 4 (+2) 1.3 mg/m2 on days 1 and 4
Period: Overall Study
Arm/Group | Arm 1
Started | 76
Completed | 76
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Untreated DLBCL: with untreated Diffuse Large B-cell Lymphoma (n = 40)
- Untreated MCL: with untreated mantle cell Non-Hodgkin's Lymphoma
- Total: Total of all reporting groups
Arm/Group | Untreated DLBCL | Untreated MCL | Total
Number analyzed (Participants) | 40 | 36 | 76
Age, Continuous [Median (Full Range); unit: years] | 56 [20 to 87] | 66 [45 to 80] | 63 [20 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 6 | 19
  Male | 27 | 30 | 57

OUTCOME MEASURES:

1. Primary Outcome: ORR
Description: Overall Response Rate
Time Frame: 6 cycles (18 weeks)
Measure: Number; unit: percentage of patients
Arm/Group | Untreated DLBCL | Untreated MCL
Number analyzed (Participants) | 40 | 36
percentage of patients | 88 | 81

ADVERSE EVENTS:
Arm/Group | Arm 1
Serious Adverse Events (participants affected / at risk) | 1/76
Other Adverse Events (participants affected / at risk) | 76/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=76)
Uroepithelial carcinoma (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 (N=76)
Neutropenia (Blood and lymphatic system disorders) | 42 — Neutropenia
Anemia (Blood and lymphatic system disorders) | 60 — Anemia
Thrombocytopenia (Blood and lymphatic system disorders) | 59 — Thrombocytopenia
Febrile Neutropenia (Infections and infestations) | 13 — Febrile Neutropenia
Infection (normal ANC) (Infections and infestations) | 14 — Infection (normal ANC)
Sepsis (Infections and infestations) | 6 — Sepsis
Neuropathy (Nervous system disorders) | 49 — Neuropathy
Anorexia (Gastrointestinal disorders) | 31 — Anorexia
Nausea (General disorders) | 33 — Nausea
Constipation (Gastrointestinal disorders) | 37 — Constipation
Diarrhea (Gastrointestinal disorders) | 25 — Diarrhea
Edema (General disorders) | 18 — Edema
Vomiting (General disorders) | 14 — Vomiting
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 18 — Dyspnea
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 — Pleural effusion
Interstitial pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 — Interstitial pneumonitis
Cardiac Arrhythmia (Cardiac disorders) | 6 — Cardiac Arrhythmia
Congestive heart failure (Cardiac disorders) | 2 — Congestive heart failure
acute renal failure (Renal and urinary disorders) | 2 — acute renal failure
Deep Vein Thrombosis (Blood and lymphatic system disorders) | 2 — Deep Vein Thrombosis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes